CLINICAL TRIAL: NCT04029233
Title: Prospective, Open-label, Multicenter, Non-randomized Investigation on Percutaneous Patent Foramen Ovale (PFO) Closure Using the Occlutech PFO Occluder to Prevent Recurrence of Stroke in Patients With Cryptogenic Stroke and High Risk PFO
Brief Title: The PROOF Trial - Prospective, Open-label, Multicenter, Non-randomized Investigation on Percutaneous Patent Foramen Ovale (PFO) Closure Using the Occlutech PFO Occluder to Prevent Recurrence of Stroke in Patients With Cryptogenic Stroke and High Risk PFO
Acronym: PROOF
Status: Terminated | Type: Observational
Why Stopped: Not due to safety concerns,high procedure success rate,6mo closure rate 94.2%,rate of SADE1.1%, 12mo rcurrent stroke rate 0.8%.Concurrent OCCLUFLEX trial+projected completion earlier than PROOF FU,no need to demonstrate add.level of efficacy evidence
Sponsor: Occlutech International AB (Industry)
Responsible Party: Sponsor
Other Study IDs: Occ2019_01
Record Dates: First submitted 2019-07-18; First posted 2019-07-23 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Stroke; PFO - Patent Foramen Ovale
MeSH Terms: conditions — Stroke; Foramen Ovale, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Occlutech PFO Occluder — The Occlutech PFO Occluder is a medical device for transcatheter closure of PFO.
  Other Names: Occlutech Figulla Flex II Occluder

SUMMARY:
Percutaneous transcatheter closure of a patent foramen ovale (PFO) to reduce the risk of recurrent ischemic stroke in patients who have had a cryptogenic stroke due to a presumed paradoxical embolism.

DETAILED DESCRIPTION:
This study aims to investigate stroke recurrence rates after interventional PFO closure with an Occlutech PFO Occluder in patients who have experienced at least one ischemic cryptogenic stroke attributed to patent foramen ovale (PFO) who have high risk PFO, i.e. large PFO (≥2 mm), or PFO of any size and atrial septal aneurysm (ASA).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years and ≤65 years
* At least one event of cryptogenic ischemic stroke in the last 12 months
* Presence of a PFO indicated for device-assisted closure (in compliance with the Instruction for Use) confirmed by common practice procedures
* A large PFO (maximum separation of the septum primum from the secundum) of ≥2 mm confirmed by common practice procedures, or an ASA defined by common practice procedures as septum primum excursion of ≥10 mm
* Life expectancy of at least 1 year
* Ability to speak fluently and to understand the language in which the study is being conducted
* Written, informed consent by the patient for participation in the study and agreement to comply with the follow-up schedule

Exclusion Criteria:

* Acute infection(s)
* Known coagulation disorder
* Arrhythmia
* Atrial Tumor
* Allergies to nickel and/or titanium and/or nickel/titanium-related material
* Inability to achieve adequate oral anticoagulation therapy and/or platelet inhibition post intervention
* Intolerance to contrast agents
* Participation in another clinical investigation <30 days before intended Occlutech PFO Occluder implantation procedure (note that in line with Medical Device Reporting, registries are not considered as clinical investigations)
* Contraindication to use of trans-esophageal echocardiography (TEE) and/or use of general anesthetic
* Eisenmenger Syndrome
* Recent pelvic venous thrombosis
* Myocardial infarction or coronary artery bypass surgery within the last 30 days
* Atrial thrombus
* Patients whose size or condition would cause them to be a poor candidate for cardiac catheterization (e.g. too small for echocardiography imaging probe, catheter size, vasculature size, active infection, body weight <8 kg)

The following exclusion criteria are at the discretion of the investigator:

* Stroke of any other origin
* Large artery atherosclerosis
* Small vessel disease
* Arterial dissection
* Hypercoagulable disorder
* Uncontrolled hypertension
* Uncontrolled diabetes
* Autoimmune disease
* Evidence of drug or alcohol abuse
* Chronic, persistent, or paroxysmal atrial fibrillation or atrial flutter
* End-stage heart-, liver-, lung-, or kidney disease
* Cardiac tumor
* Endocarditis or septicemia
* Severe valvular pathology
* Any condition that, in the opinion of the investigator, might interfere with the implantation,might affect the patients' well-being thereafter or might interfere with the conduct of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will enroll patients of either sex, aged ≥18 and ≤60 years, with at least one event of cryptogenic ischemic stroke in the last 6 months. Patients must have a high risk PFO indicated for device-assisted closure; either large PFO (≥2 mm), or PFO of any size and ASA.
Sampling Method: Probability Sample
Enrollment: 582 (Actual)
Dates: Start 2019-10-03 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
To demonstrate the safety and tolerability of the Occlutech PFO occluder by assesssing the incidence of SADEs. | in the 1 year following implantation.
To demonstrate the medium-term effectiveness of the Occlutech PFO Occluder by assessing the rate of ischemic strokes. | in the 5 years following implantation

CONTACTS AND LOCATIONS:
Locations (17):
- St. Paul's Hospital, Vancouver, Canada
- France (4):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - Institut de Cardiologie,groupe hospitalier pitié salpêtrière, Paris
  - New Civil Hospital, Strasbourg
  - CHU Rangueil, Toulouse
- Germany (11):
  - Charité Universität Berlin, Berlin
  - Herzzentrum Bremen, Bremen
  - Klinikum Coburg, Coburg
  - Herzzentrum der Universität zu Köln, Cologne
  - Herzzentrum Dresden Universitätsklinik an der Technischen Universität Dresden, Dresden
  - Universitätsklinikum Düsseldorf, Düsseldorf
  - CardioVasculäres Centrum Frankfurt, Frankfurt
  - Uniklinik Freiburg, Freiburg im Breisgau
  - Asklepios Klinik Hamburg, Hamburg
  - Uniklinik Heidelberg, Heidelberg
  - University Jena, Jena
- Centro Cardiologico Monzino, Milan, Italy